CLINICAL TRIAL: NCT06680778
Title: The Use of Proa-active Monitoring by Measuring Vital Signs Using a Fitbit for a 3-month Period Before, During, and After Chemotherapy in Patients With Cancer
Brief Title: Pro-active Monitoring of Vital Signs in Oncology Patients Using a Smartwatch
Acronym: PROGRESS
Status: Recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Jason den Duijn, Principal Investigator, Erasmus Medical Center
Other Study IDs: 13016
Record Dates: First submitted 2024-10-14; First posted 2024-11-08 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Cancer; Emergencies
Keywords: cancer; monitoring; Fitbit
MeSH Terms: conditions — Neoplasms; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cancer Patients: All patients with stomach and esophageal malignancies referred for chemotherapy of the outpatient clinic at the department of Medical Oncology at the Erasmus University Medical Center.
  Interventions: Device: Proactive Monitoring

INTERVENTIONS:
Device: Proactive Monitoring — Proactive monitoring of vital signs for the duration of the first two cycles of chemotherapy by using a Fitbit

SUMMARY:
The goal of this single center prospective observational study is to determine the effect of chemotherapy on (the change in) vital parameters. The main question it aims to answer are: Can changes in vital parameters be measured by using a Fitbit in patients with cancer while undergoing chemotherapy. Participants will be asked to wear a Fitbit for the first two cycles of chemotherapy to evaluate the changes in vital parameters.

DETAILED DESCRIPTION:
The goal of this single center prospective observational study is to determine the effect of chemotherapy on (the change in) vital parameters. The main question it aims to answer are: Can changes in vital parameters be measured by using a Fitbit in patients with cancer while undergoing chemotherapy. Participants will be asked to wear a Fitbit for the first two cycles of chemotherapy to evaluate the changes in vital parameters. Patients will start measuring in the week prior to the first cycle of chemotherapy, target is at least 4 to 7 days before initiation of chemotherapy. Patients were the Fitbit as much as possible, during day and night. Patients continuously carry the Fitbit during the first 3 months of systemic treatment, which tracks their vital signs. At the starting day of the next cycle of chemotherapy patients will have an appointment with one of the researchers to evaluate the use of the Fitbit. Furthermore, it will be checked if a patient has returned to their baseline vital signs.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Diagnosis of stomach or esophageal cancer with an indication of starting chemotherapy
* Knowledge how to handle a Fitbit
* Mastery of Dutch language
* Able and willing to give written informed consent

Exclusion Criteria:

* Cognitive disorders or severe emotional instability
* Already participating in an exercise trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with stomach and esophageal malignancies referred for chemotherapy of the outpatient clinic at the department of Medical Oncology at the Erasmus University Medical Center.
Sampling Method: Probability Sample
Enrollment: 175 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Variance and normalization of resting heart rate | Through study completion, an average of 6 months
  Variance and normalization of resting heart rate in bpm over time during chemotherapy
Variance and normalisation of maximum heart rate | Through study completion, an average of 6 months
  Variance and normalization of vital parameters maximum heart rate in bpm over time during chemotherapy
Variance and normalisation of minimum heart rate | Through study completion, an average of 6 months
  Variance and normalization of minimum heart rate in bpm over time during chemotherapy
Variance and normalisation of heart rate variability | Through study completion, an average of 6 months
  Variance and normalization of vital parameters heart rate variability over time during chemotherapy
Variance and normalisation of respiratory rate | Through study completion, an average of 6 months
  Variance and normalization of respiratory rate in absolute numbers over time during chemotherapy
Variance and normalisation of blood pressure | Through study completion, an average of 6 months
  Variance and normalization of blood pressure in mmHG over time during chemotherapy
Variance and normalisation of step count | Through study completion, an average of 6 months
  Variance and normalization of step count in absolute numbers over time during chemotherapy
Variance and normalisation of blood oxygen saturation | Through study completion, an average of 6 months
  Variance and normalization of blood oxygen saturation in percentage over time during chemotherapy
Variance and normalisation of sleep time | Through study completion, an average of 6 months
  Variance and normalization of sleep time in hours over time during chemotherapy
Variance and normalisation of sleep quality | Through study completion, an average of 6 months
  Variance and normalization of sleep quality on a scale from 1 to 10 over time during chemotherapy

SECONDARY OUTCOMES:
Contact with healthcare provider | Through study completion, an average of 6 months
  Number of contact moments with a healthcare provider (nurse, nurse practioner, general practioner, treating physician)
emergency department visits | Through study completion, an average of 6 months
  Number of emergency department visits
Toxicity | Through study completion, an average of 6 months
  Toxicity, defined as a grade between 1 and 4, documented in electronic patient file
Dose Modification of chemotherapy | Through study completion, an average of 6 months
  Modification in dosage of chemotherapy, documented in electronic patient file

OTHER OUTCOMES:
Age group | Through study completion, an average of 6 months
  Group (18-30, 31-50, 51-65, 65+) of age of participant
Sex | Through study completion, an average of 6 months
  Sex (male/female) of patient
Cancer Type | Through study completion, an average of 6 months
  The cancer diagnosis of the patient
Type of Chemotherapy | Through study completion, an average of 6 months
  The specific chemotherapy a patient will receive

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus University Medical Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No